CLINICAL TRIAL: NCT00005629
Title: Phase I/II Trial Testing Alpha Fetoprotein (AFP) Peptide Immunization in Hepatocellular Carcinoma
Brief Title: Vaccine Therapy in Treating Patients With Liver Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: James Economou, MD / Principal Investigator, UCLA
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067782; UCLA-9905003; NCI-H00-0053
Record Dates: First submitted 2000-05-02; First posted 2003-10-01 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Liver Cancer
Keywords: localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A - first dosing group (Experimental): Patients will receive three biweekly intradermal vaccinations with four HLA-A*0201-binding AFP-derived peptides (100 ug dose) emulsified in 2 ml of Montanide ISA-51.
  Interventions: Biological: AFP gene hepatocellular carcinoma vaccine
- Arm B - dosing group 2 (Experimental): Patients will receive three biweekly intradermal vaccinations with four HLA-A*0201-binding AFP-derived peptides (500 ug dose) emulsified in 2 ml of Montanide ISA-51.
  Interventions: Biological: AFP gene hepatocellular carcinoma vaccine
- Group 3 - dosing level 3 (Experimental): Patients will receive three biweekly intradermal vaccinations with four HLA-A*0201-binding AFP-derived peptides (1000 ug dose) emulsified in 2 ml of Montanide ISA-51.
  Interventions: Biological: AFP gene hepatocellular carcinoma vaccine

INTERVENTIONS:
Biological: AFP gene hepatocellular carcinoma vaccine — Patients will receive three biweekly intradermal vaccinations with four HLA-A*0201-binding AFP-derived peptides emulsified in 2 ml of Montanide ISA-51.
  Group A AFP peptide dose 100 ug Group B AFP peptide dose 500 ug Group C AFP peptide dose 1000 ug

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of vaccine therapy in treating patients who have liver cancer.

ELIGIBILITY:
Inclusion Criteria

* This study will enroll HLA-A 0201 adults over the age of 18 with history of biopsy-proven HCC and AFP positive by immunohistochemistry or serum AFP levels > 2 times above the upper limit of normality. Any stage of disease will be eligible.
* Both male and female patients may be enrolled. Females of childbearing potential must have a negative pregnancy test prior to treatment.
* Patients must be ambulatory with a Karnofsky Performance Status greater than or equal to 70 percent.
* No previous evidence of class 3 or greater New York Heart Association cardiac insufficiency or coronary artery disease.
* No evidence of opportunistic infection.
* A minimum of 4 weeks must have elapsed since the completion of prior chemotherapy or radiation therapy.
* Adequate baseline hematological function as assessed by the following laboratory values within 30 days prior to study entry (day -30 to 0):

  * Hemoglobin > 8.5 g/dl (patients cannot be transfusion dependent).
  * Platelets > 30,000/mm3
  * WBC > 2,000/mm3
  * Absolute Neutrophil Count (ANC) > 1,000/mm3
* Positive skin test to common antigens (tetanus and/or candida).
* Ability to give informed consent and signed informed consent.

Exclusion Criteria

Patients who meet any one of the following criteria will be excluded from study entry:

* Any congenital or acquired condition leading to inability to generate an immune response, including concomitant immune suppressive therapy. The ability to adequately respond to antigens will be tested before trial entry by requiring a positive response to skin allergens (tetanus and candida).
* Lactating females: All patients must practice adequate birth control and females of child-bearing potential must have a negative serum HCG pregnancy test (within day -7 to day 0).
* Acute infection: any acute viral, bacterial, or fungal infection, which requires specific therapy. Acute therapy must have been completed within 14 days prior to study treatment.
* HIV-infected patients, due to concerns in the ability to stimulate an effective immune response.
* Acute medical problems such as ischemic heart or lung disease that may be considered an unacceptable anesthetic or operative risk.
* Patients with any underlying conditions that would contraindicate therapy with study treatment (or allergies to reagents used in this study).
* Patients with organ allografts.
* Uncontrolled hepatic insufficiency and cirrhosis, Class C in the Child's classification, with bilirubin > 3 mg/dl, albumin < 3.0 g/dl, poorly controlled ascites, advanced encephalopathy and poor nutritional status.
* Uncontrolled CNS metastasis. Patients with previously known CNS metastasis will be eligible if they have received CNS irradiation to control local tumor growth.
* Concomitant Medication and Treatment:

All allowed medications or treatments should be kept to a minimum and recorded.

- Concomitant Medications and Treatments Not Allowed: Corticosteroids, Cyclosporin A, cytotoxic chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1999-07; Primary Completion 2002-05 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Safety | 1 month
  Determine the safety of intradermal injection of the hAFP137-145 (PLFQVPEPV), hAFP158-166 (FMNKFIYEI), hAFP325-334 (GLSPNLNRFL) and hAFP542-550 (GVALQTMKQ) peptides emulsified in Montanide ISA-51.

SECONDARY OUTCOMES:
antigen-specific immune response | 1 month
  Determine the antigen-specific immune response to hAFP137-145 (PLFQVPEPV), hAFP158-166 (FMNKFIYEI), hAFP325-334 (GLSPNLNRFL) and hAFP542-550 (GVALQTMKQ), emulsified with Montanide ISA-51, in peripheral blood of patients with liver cancer.
Survival | 1 month
  Determine the overall survival, disease-free survival or progression-free survival of patients with HCC vaccinated with hAFP137-145 (PLFQVPEPV), hAFP158-166 (FMNKFIYEI), hAFP325-334 (GLSPNLNRFL) and hAFP542-550 (GVALQTMKQ), emulsified with Montanide ISA-51.

CONTACTS AND LOCATIONS:
Overall Officials: James S. Economou, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States